CLINICAL TRIAL: NCT00055341
Title: A Prospective Multicenter, Phase II, Open Label, Controlled Trial Evaluating the Response of Hepatitis C Virus (HCV) to Pegylated Interferon Alpha-2A and Ribavirin in Hemophilic Patients With and Without Coinfection With the Human Immunodeficiency Virus (HIV)
Brief Title: Treatment of Hepatitis C in Hemophilic Patients With HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R01AI049508-01 (NIH); 5R01AI049508-02 (NIH)
Record Dates: First submitted 2003-02-25; First posted 2003-02-27 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2006-12

CONDITIONS: HIV Infections; Hepatitis C; Hemophilia
MeSH Terms: conditions — HIV Infections; Hepatitis C; Hemophilia A | interventions — peginterferon alfa-2a; Ribavirin

INTERVENTIONS:
Drug: Peginterferon alfa-2a
Drug: Ribavirin

SUMMARY:
Pegylated interferon (PEG-interferon) and ribavirin are accepted treatments for hepatitis C virus (HCV) infection. However, HCV infection progresses differently in patients who are coinfected with HIV and in hemophiliacs. This study will evaluate the effectiveness of PEG-interferon and ribavirin for treating HCV in HIV infected hemophiliacs.

DETAILED DESCRIPTION:
Hemophiliacs with symptomatic disease often receive blood products to correct clotting factor deficiencies. Prior to routine use of heat inactivation and screening of donor blood for specific viral pathogens, hemophiliacs were routinely exposed to, and infected with, viruses such as hepatitis B (HBV), HCV, and HIV. Studies in hemophiliacs suggest several important findings that warrant further investigation, including: 1) hemophiliacs infected with HCV may have more rapid progression to liver failure and death; 2) pooled blood concentrate from multiple donors leads to a high risk of mixed infection; and 3) different clinical outcomes and altered immune responses of HIV coinfected hemophiliacs may enhance understanding of mutant virus selection and the associated clinical outcomes. The purpose of this trial is to determine response rates to PEG-interferon and ribavirin in hemophiliacs with HCV alone and with HCV/HIV coinfection.

Participants in this study will be followed for 48 weeks on treatment and up to 36 months after treatment. Participants in this study will be admitted to the Clinical Research Center for 2 days at the beginning of the study. Participants will have 3 additional study visits in the first week of the study. After that, study visits occur at Weeks 2, 4, 8, 12, 16, 24, 32, 40, and 48. The follow-up visits will be at 4, 12, and 24 weeks following the end of treatment. Study visits include a physical exam and blood tests. Patients who do not respond to treatment will be followed in a prospective cohort study for up to 3 additional years so that evolution of the virus and associated immune responses can be evaluated.

ELIGIBILITY:
Inclusion Criteria

* Hemophilia A or B
* Exposure to blood or blood products prior to 1987
* Participating in "The Second Multicenter Hemophilia Cohort Study (MHCS-II)"
* HCV reactive by second/third generation ELISA assay and/or RIBA
* HCV RNA positive (PCR or bDNA methods)
* Chronic hepatitis confirmed by liver biopsy within 6 months prior to study entry (Note: cirrhosis is not an exclusion factor)
* HIV infection for coinfected group; HIV viral load of 10,000 copies/ml or less
* If on antiretroviral drugs, stable regimen for at least 8 weeks prior to study entry
* Acceptable methods of contraception

Exclusion Criteria

* Hemoglobin less than 10 g/dl
* For HIV coinfected group, CD4 count less than 200 cells/mm3 at time of screening visit
* Previous interferon or ribavirin therapy
* Corticosteroids or immunomodulatory drugs within 3 months prior to study entry
* Hepatitis B (HBsAg reactive)
* Alpha-1 antitrypsin deficiency
* Wilson's disease
* Hemochromatosis
* Autoimmune disorder
* Decompensated liver disease evidenced by encephalopathy, ascites, or variceal bleed
* Prothrombin Time greater than 3 seconds above normal (International Normalized Ratio [INR] greater than 1.3)
* Platelet count less than 90,000/microL
* Active thyroid disease (thyroid replacement with normal TSH permitted)
* Chronic renal insufficiency, defined as creatinine greater than 1.5 mg/dl
* Life-threatening disease processes that could preclude completion of trial
* Alcohol abuse that the local investigator feels would interfere with compliance
* Illicit recreational drug use or methadone use within 6 months of study entry
* Major depression with hospitalization or suicide attempt is a relative, but not absolute, contraindication to therapy based on timing, circumstances, and current stability as assessed by the investigator
* Pregnant or breastfeeding

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22
Dates: Start 2002-03; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth E. Sherman, MD, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Result] Shire NJ, Horn PS, Rouster SD, Stanford S, Eyster ME, Sherman KE; Multicenter Hemophilia Cohort HCV Study Group. HCV kinetics, quasispecies, and clearance in treated HCV-infected and HCV/HIV-1-coinfected patients with hemophilia. Hepatology. 2006 Nov;44(5):1146-57. doi: 10.1002/hep.21374. PMID 17058240
- [Result] Qin H, Shire NJ, Keenan ED, Rouster SD, Eyster ME, Goedert JJ, Koziel MJ, Sherman KE; Multicenter Hemophilia Cohort Study Group. HCV quasispecies evolution: association with progression to end-stage liver disease in hemophiliacs infected with HCV or HCV/HIV. Blood. 2005 Jan 15;105(2):533-41. doi: 10.1182/blood-2004-04-1452. Epub 2004 Sep 16. PMID 15374882